CLINICAL TRIAL: NCT06123078
Title: Impact of Schemas, Cognitive Emotion Regulation on Quality of Life of HIV Patients: Assessing Outcomes of CBT
Acronym: Step-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Islamia University of Bahawalpur (Other)
Responsible Party: Principal Investigator, Rabia Javed Bhatti, Principal Investigator, Islamia University of Bahawalpur
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 123987
Record Dates: First submitted 2023-10-14; First posted 2023-11-08 (Actual); Last update posted 2023-11-08 (Actual); Status verified 2023-11

CONDITIONS: Quality of Life

STUDY DESIGN:
Intervention Model Description: Repeated measures design
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double blind control technique
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): treatment as usual
- Experimental group (Experimental): CaCBT
  Interventions: Behavioral: CaCBT

INTERVENTIONS:
Behavioral: CaCBT — Culturally adapted Self help guide and modules total eight 80 hour session per week
  Arms: Experimental group

SUMMARY:
The present study has investigated the impact of schemas, cognitive emotion regulation and social connectedness on the Quality of life of HIV patients in South Punjab region, Pakistan.

DETAILED DESCRIPTION:
The present study has investigated the impact of schemas, cognitive emotion regulation and social connectedness on the Quality of life of HIV patients in South Punjab region, Pakistan. The main study was conducted in four steps as follows:

Step 1: Pre-testing, N=150 Baseline assessment Random assignment of willing participants to control and experimental Step 2: CBT Intervention, N=40, 20 each group Step 3: post-test Step 4: Follow up Assessmen

ELIGIBILITY:
Inclusion Criteria:

- Registered at ART clinics South Punjab region HIV Patients Stage 1 or stage 2 Understands urdu Age above 20

Exclusion Criteria:

AIDS converted No Other terminal illness No other diagnosis Below 20 age

Ages: 20 Years to 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Male
Enrollment: 40 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Social Connectedness Scale SCS-R | 8 months
  To measure social connectedness
WHOQOL-HIV Bref | 8 months
  HiV patients Quality of life will be enhanced
Schema Mode Inventory | 8 months
  This helped to measure schemas
CERQ | 8 months
  To measure cognitive emotion regulation strategies
WHOQOL | 8 months
  After intervention on HIV patients, Quality of Life will be enhanced as an outcome of the CBT intervention

OTHER OUTCOMES:
Cognitive Behavioural therapy | 4 months
  CBT Intervention will be given to HIV patients

CONTACTS AND LOCATIONS:
Overall Officials: Rabia J Bhatti, PhD, Principal Investigator — The Islamia University of Bhawalpur
Locations (2):
- Pakistan (2):
  - Nai Zindagi Trust, Rahim Yar Khan, Punjab Province
  - Sheikh Zyed Hospital, Rahim Yar Khan, Punjab Province

IPD SHARING:
Plan to Share IPD: No
Data is sensitive, can assess directly by the principle investigator